CLINICAL TRIAL: NCT04271813
Title: Anlotinib Plus Sintilimab as First-line Treatment for Patients With Advanced Colorectal Cancer (APICAL-CRC): a Single Center, Single-arm Phase II Study (APICAL-CRC)
Brief Title: Anlotinib Plus Sintilimab as First-line Treatment for Patients With Advanced Colorectal Cancer (APICAL-CRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Director, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APICAL-CRC
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Immunotherapy; Anlotinib; Sintilimab; Chemo-free Therapy; First-line Treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib and Sintilimab (Experimental): the combination of Anlotinib with Sintilimab as first-line treatment
  Interventions: Drug: Anlotinib plus Sintilimab

INTERVENTIONS:
Drug: Anlotinib plus Sintilimab — Anlotinib 12mg oral administration daily d1-d14, q3w; Sintilimab 200mg iv drop d1, q3w

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination of Anlotinib and Sintilimab in advanced colorectal cancer as first-line treatment.

DETAILED DESCRIPTION:
Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR), and c-kit. Sintilimab is a fully human IgG4 monoclonal antibody that binds to programmed cell death receptor-1 (PD-1), thereby blocking the interaction of PD-1 with its ligands (PD-L1 and PL-L2) and consequently helping to restore the endogenous antitumour T-cell response. In the present study, we design a single-arm, single center Phase II trial to evaluate the efficacy and safety of the combination of Anlotinib and Sintilimab in advanced colorectal cancer as first-line treatment.

ELIGIBILITY:
Inclusion criteria

* Patients have histologically or cytologically confirmed advanced or recurrent CRC;
* No prior systematic anti-cancer treatment and relapse or metastases was occurred more than 12 months after adjuvant chemotherapy;
* Patients have measurable disease as defined by RECIST 1.1 as determined by investigator;
* Patient with a history of radiotherapy at least 3 months before on the day of providing consent, but the measurable lesion should not be within the scope of radiotherapy;
* Patients with age of 18-75yr;
* Patients with a performance status of 0,1or 2 on the Eastern Cooperative Oncology Group.；
* Patients with Life expectancy of more than 12 weeks;
* Patients must have the ability to understand and sign the written informed consent voluntarily;
* Female of childbearing potential who are negative in a pregnancy test within 7 days before enrollment. Both male and female patients should agree to use an adequate method of contraception (total abstinence, an intrauterine device or hormone releasing system, a contraceptive implant and an oral contraceptive) starting with the first dose of study therapy through 120 days after the last dose of study therapy. Duration will be determined when the subject is assigned to treatment.

Exclusion criteria

* Patients with dMMR/MSI-H;
* Patients with major surgery or severe trauma within 4 weeks before the first medication;
* Patients with hypersensitivity to the components in the study protocol;；
* Patients who are ready to give birth or are pregnant;
* Patients with brain metastases who are unable to accurately describe the condition;
* Patients received immune-suppressive drugs 2 weeks before initial treatment (inhaled cortisol or other steroid hormones≤10 mg/day prednisone or equivalent pharmacophysiologic doses were excluded);
* Planned live attenuated vaccine within 4 weeks prior to or during study treatment;
* Patients have received anlotinib or anti-PD-1 monoclonal antibody therapy or other therapies that act on T-cell co-stimulation targets or checkpoints;
* Within 6 months prior to the start of study treatment, the following diseases appeared: myocardial infarction, severe/unstable angina, NYHA grade 2 or above congestive heart failure, poorly controlled arrhythmias, etc;
* Active hepatitis;
* Bone marrow, liver and kidney function did not meet the requirements of chemotherapy as follows:

  * Neutrophil count<1,500/mm3;
  * Platelet count <80,000/mm3;
  * Total bilirubin >1.5-times the upper limit of normal;
  * ALT/AST>2.5-times the upper limit of normal for patients without liver metastases; (5.0-times the upper limit of normal for patients with liver metastases)
  * Creatinine >1.5-times the upper limit of normal;
* Patients with cancers other than advanced colorectal cancer within five years prior to the start of treatment in this study. Cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor were excluded;
* History of substance abuse, drug use, alcohol dependence;
* Patients without legal capacity or limited civil capacity;
* Patients with autoimmune diseases or organ transplantation;
* Other situations that the investigator deemed inappropriate for enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Objecitve response rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 6 weeks
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

SECONDARY OUTCOMES:
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 6 weeks
  Time from treatment beginning until disease progression
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 3 weeks
  Time from treatment beginning until death from any cause
Incidence of Treatment-related adverse Events | Through study completion, an average of 3 weeks
Deepness of response | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 6 weeks
  Investigation of depth of response during first-line treatment
Disease control rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 6 weeks
  Proportion of patients who achieved a complete response, a partial response, or stable diseas

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Qin BD, Ye CY, Wang MM, Yuan LY, Yao HS, Jiao XD, Liu K, Zhou WL, Qin WX, Sun L, Dai WP, Ling Y, Wu Y, Chen SQ, Zhang YF, Shi DM, Duan XP, Zhong X, He X, Zhai WX, Zhang B, Zhang DD, Gao N, Zang YS. Anlotinib plus sintilimab as first-line treatment for patients with advanced colorectal cancer (APICAL-CRC): an open-label, single-arm, phase II trial. Signal Transduct Target Ther. 2025 Sep 16;10(1):301. doi: 10.1038/s41392-025-02383-9. PMID 40954146